CLINICAL TRIAL: NCT01439269
Title: Enhancement of Co-regulation Between Mother and Infant Via Family Nurture Intervention (FNI) in the NICU: Short and Long Term Effects on Development
Brief Title: Family Nurture Intervention (FNI) in Neonatal Intensive Care Unit (NICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Williams College (Other); New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Martha G Welch, Assistant Professor of Clinical Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAD0389
Record Dates: First submitted 2011-09-19; First posted 2011-09-23 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Premature Birth
Keywords: Separation stress; Family Nurture; Maternal Confidence; Maternal Competence; Calming Cycle; Kangaroo Care; Infant Neurodevelopment; Infant Psychological Development; Post-partum depression; Mother-infant Co-regulation
MeSH Terms: conditions — Premature Birth; Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1: Standard Care (No Intervention): Mothers are given infant care instruction as part of standard care
- Phase 1: Facilitated infant care (Experimental): Family Nurture Intervention (FNI)
  Interventions: Behavioral: Family Nurture Intervention
- Phase 2: Effectiveness (Active Comparator): All participants receiving FNI
  Interventions: Behavioral: Family Nurture Intervention

INTERVENTIONS:
Behavioral: Family Nurture Intervention — Family Nurture Intervention is facilitated by specially trained Nurture Specialists. The intervention involves calming interactions between mother and infant in the isolette via odor exchange, firm sustained touch and vocal soothing, through calming interactions during holding and feeding via the Calming Cycle and through family sessions designed to engage the help and support of family members for the mother.
  Arms: Phase 1: Facilitated infant care; Phase 2: Effectiveness

SUMMARY:
The purpose of this study is to test the efficacy of a family nurture intervention in the neonatal intensive care unit (NICU). Infants receiving enhanced mother-infant and family nurture are compared to infants receiving standard NICU care. The intervention enhances mother/infant interactions that are vital to early development in the infant. The main goal is to get the mother and infant into biological synchrony, emotional attunement and mutual calm through an activity referred to as a "calming cycle". Mother's are encouraged to engage in the calming cycle activities as much as possible. Her increased effectiveness in calming her infant is hypothesized to improve the mother's view of her baby, reduce negative emotions about having delivered a baby prematurely, and help her gain confidence in her care-taking abilities, which in other studies predicted shorter length of stay and fewer re-hospitalizations. Another goal is to assist mothers in repeating the calming cycle activities providing appropriate types of stimulation for their babies that are important for social, emotional, and neurobehavioral development. Since preterm babies are often easily upset, mothers will be taught how to comfort and calm their babies. Assessments in the NICU and in follow-up visits for two years will test the immediate and long-term effects of this new approach to the nurture of prematurely born infants.

DETAILED DESCRIPTION:
The stress that results from preterm birth, requisite acute care and prolonged physical separation in the NICU can have adverse physiological/psychological effects on both the infant and the mother. In particular, the experience compromises the establishment and maintenance of an optimal mother-infant relationship. Within the neonatal intensive care unit (NICU), parental involvement in care is necessarily superseded by the healthcare staff. Thus, a necessary but detrimental separation between mother and infant is created at a critical period when mother-infant bonding and synchrony should be developing. The physiological challenges associated with being born too soon, along with disturbances in normal mother-infant interactions are key factors underlying the risks of premature infants for a broad range of early and midlife disorders. This study aims to highlight the importance of investigating early interventions that are designed to overcome or reduce the effects of these environmental insults and challenges by implementing a randomized controlled trial of Family Nurture Intervention in the NICU. The most important source of regulatory input is through contact with the mother and her nurturing behavior. Mother-infant interactions are the foundation for the organization of the infant's neurobiological, sensory, perceptual, emotional, physical, and relational systems. The infant's responses to the mother provide critical feedback which shapes her behavior as well. There are many co-regulatory processes embedded in these synchronous and reciprocal interactions which cross neurophysiological and neurobehavioral domains. The intervention is designed to increase biologically important activities and behaviors that enhance maternally-mediated sensory experiences of preterm infants, as well as the infant-mediated sensory experiences in the mother. The investigators hypothesize that repeated engagement of the mother and her infant in the intervention's calming activities will increase the effectiveness of co-regulation and have immediate and long-term beneficial effects for both. The study is assessing the physiological and behavioral outcomes of the infants and mothers receiving Family Nurture Intervention versus Standard Care over the course of the NICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Infant is born a singleton or twin in the Morgan Stanley Children's Hospital in New York City
* Infant is born 26 and 34 weeks post-conceptional age (PCA)

Exclusion Criteria:

* Mothers cannot understand or speak English
* Mother has history of drug addiction, psychosis or other severe mental illness
* There is not at least one adult other than the mother in the home
* Infant birth weight is below the third percentile for gestational age
* Infant has significant congenital defects

Ages: 26 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 394 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2012-07-03 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Length of Stay | From Infant's birth to discharge from NICU
  Length of stay will be determined based on the infant's number of days as an inpatient at the Children's Hospital of New York (CHONY) NICU.

SECONDARY OUTCOMES:
Safety and Practicability of Intervention | up to 5 years
  To confirm implementation of the intervention is safe and practicable within the Neonatal Intensive Care Unit (NICU)throughout the study duration.
Psychological Assessments: Mothers in both groups are given a wide-range of psychological questionnaires. These include indices of anxiety, depression, temperament, personality, attachment, stress, and social support. | Up to 24 months of Age
  Mothers are administered questionnaires at several time periods to assess levels of anxiety (Speilberger State-Trait Anxiety Inventory), and depressive symptoms (Center for Epidemiological Studies Depression Scale). After group assignment, symptoms of post-partum depression (Postpartum Depression Screening Scale), depressive experiences (Depressive Experiences Questionnaire), qualities of attachments (Adult Attachment Interview) are assessed. Status of inhibitory vs. approach systems (Behavioral Inhibition System-Behavioral Approach System), and Mom's Support Circle are assessed.
Neurobehavioral Assessments of Infants: The use of the NICU Network Neurobehavioral Scale (NNNS) to assess infant's neurodevelopmental status | Up to 40 weeks Gestational Age
  The test measures neurological reflexes, body tone and motor maturity at 36 weeks (+/- 1 week) and 40 weeks (+/- 1 week) post-conceptional age. It also measures the infant's orientation to and engagement with social and non-social stimuli, the lability of the infant's activity and states, and the infant's consolability. The stress/abstinence scale, originally formulated for prenatally drug-exposed infants, includes physiological, autonomic, skin, central nervous system (CNS), visual and gastrointestinal markers.
Neurobehavioral Assessments of Infants: Mothers provide a wide range of information about infant's development through questionnaires | Up to 24 months corrected age
  Infant temperament is obtained using the Early Infancy Temperament Questionnaire and the Infant Behavior Questionnaire. Social-emotional problems of the infants are assessed by the Brief Infant-Toddler Social and Emotional Assessment at 4, 12, 18 and 24 months corrected age, and at 12, 18, 24 months CA by the Child Behavior Checklist. The mother also provides information about possible developmental delays by filling out the Ages and Stages Questionnaire, at 4, 12, 18 and 24 months corrected age.
Neurobehavioral Assessments of Infants- Bayley Scales of Infant and Toddler Development, Bayley III | Up to 24 months corrected age
  At 18 and 24 months corrected age, infants are administered the Bayley Scales of Infant and Toddler Development, Bayley III consisting of four subscales: Cognitive, Language (receptive/expressive), Motor (fine/gross) and Social-Emotional. These filmed assessments, made by research staff 'blind' to infant group assignment, provide information about the neurobehavioral status of the child and whether there are significant delays in key domains of motor, language, and cognitive development.
Physiological Assessments: A one hour recording of high density electroencephalogram (EEG) (128 leads), electrocardiogram (ECG), and respiration during sleep. | Up to 42 weeks post-conceptional age
  EEG and ECG are collected at 1000 samples/sec and respiration at 50 samples/sec at 34, 36, and 39-42 weeks post-conceptional age. Throughout recording, research assistants assign sleep state codes (quiet sleep, active sleep, indeterminate, awake, cry) once each minute, based on behavioral criteria as well as provide estimates of heart rate and heart rate for each sleep state. EEG data is processed to obtain spatially-dependent measures of wave amplitude (power) at specific frequencies for each spatial location and measures of functional connectivity (coherence) between electrode locations.
Physiological Assessments- Cortisol Levels, breast milk, saliva, infant blood samples, and infant stool collection | Up to 24 months corrected age
  As a component of the mother-infant interaction assessments conducted at 4 and 12 months corrected age, salivary cortisol levels are measured at four times during each session. These measures provide physiological indices of how the infants respond to a social interaction stressor. In addition, breast milk, saliva (mother and infant), infant stool, and infant blood for peptides are collected.
Mother-Infant Interactions Assessments: Evaluating the qualities of the mother's interaction with her infant during diaper change | Up to 4 months corrected age
  Videos of infant's diaper change are obtained and coded by research team members unfamiliar with the dyads' group assignment at 36 weeks post-conceptional age and 4 months corrected age. The mother is instructed to undress her infant, remove the diaper, wipe clean, and re-dress her infant. These familiar caregiving procedures represent a mild, ecologically valid stressor. Maternal behavior is coded, using a 9-point Likert scale for: (a) Acceptance vs. Rejection; (b) Soothing capability; (c) Consideration vs. Intrusiveness; (d) Quality of Physical Contact; and (e) Quality of Vocal Contact.
Mother-Infant Interaction Assessments: Mother-infant face-to-face communicative competence, sensitivity of maternal caregiving and mother and infant physiological capacity to cope with a stressor | Up to 24 months corrected age
  A split-screen filming session is conducted following protocols and analyzed by team members 'blind' to the dyads' group assignments at 4, 12, and 24 months corrected age. The videotapes consist of: (1) mother-infant play; (2) stranger-infant play (3) diaper change; (4) the Still Face protocol in which mothers assume an expressionless face for two minutes. Primary measures are: infant gaze aversion, mother-infant gaze coordination, infant distress, maternal interaction style (affectionate vs. intrusive), and responses of mothers and infants to gaze aversion.
Mother-Infant Interaction Assessments- Yale Inventory of Parental Thoughts and Actions (YIPTA) | up to 24 months corrected age
  Twice during each infant's stay in the NICU, and again at term, 4, 12, 18 and 24 months corrected age following discharge, the Yale Inventory of Parental Thoughts and Actions, YIPTA is administered. This inventory quantifies maternal ratings of her thoughts about her infant. To evaluate the mother-to-child attachment processes subscales include: frequency of thoughts/worries about the infant, the distress caused by these thoughts, how she manages her distress, frequency of checking the infant, affiliative interactions, measures of attachment, frequency of care taking behavior.
Assessments of Neonatal Intensive Care Unit Activities: Ascertainment of attendance and the frequency and/or time spent engaged in key aspects of the Family Nurture Intervention using maternal self-report forms. | Participants will be followed for the duration of NICU stay, an expected average of 7 weeks
  These forms are filled out after each visit to NICU. The mother is asked to enter information about the start and stop times of each of her visits to the NICU and to estimate the amount of time or number of times she engaged in various types of interactions with her infant. A similar schedule of questionnaires is given to the Standard Care group mothers, but without questions that pertain only to the Family Nurture Intervention group (i.e., odor cloth exchange, Calming Cycle).

CONTACTS AND LOCATIONS:
Overall Officials: Martha G Welch, MD, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ravn IH, Smith L, Lindemann R, Smeby NA, Kyno NM, Bunch EH, Sandvik L. Effect of early intervention on social interaction between mothers and preterm infants at 12 months of age: a randomized controlled trial. Infant Behav Dev. 2011 Apr;34(2):215-25. doi: 10.1016/j.infbeh.2010.11.004. Epub 2011 Mar 2. PMID 21371754
- [Background] Muller-Nix C, Forcada-Guex M, Pierrehumbert B, Jaunin L, Borghini A, Ansermet F. Prematurity, maternal stress and mother-child interactions. Early Hum Dev. 2004 Sep;79(2):145-58. doi: 10.1016/j.earlhumdev.2004.05.002. PMID 15324994
- [Background] Meijssen D, Wolf MJ, van Bakel H, Koldewijn K, Kok J, van Baar A. Maternal attachment representations after very preterm birth and the effect of early intervention. Infant Behav Dev. 2011 Feb;34(1):72-80. doi: 10.1016/j.infbeh.2010.09.009. Epub 2010 Nov 9. PMID 21067812
- [Background] Meijssen D, Wolf MJ, Koldewijn K, Houtzager BA, van Wassenaer A, Tronick E, Kok J, van Baar A. The effect of the Infant Behavioral Assessment and Intervention Program on mother-infant interaction after very preterm birth. J Child Psychol Psychiatry. 2010 Nov;51(11):1287-95. doi: 10.1111/j.1469-7610.2010.02237.x. PMID 20345840
- [Background] Shah PE, Clements M, Poehlmann J. Maternal resolution of grief after preterm birth: implications for infant attachment security. Pediatrics. 2011 Feb;127(2):284-92. doi: 10.1542/peds.2010-1080. Epub 2011 Jan 17. PMID 21242223
- [Background] Coppola G, Cassibba R, Costantini A. What can make the difference? Premature birth and maternal sensitivity at 3 months of age: the role of attachment organization, traumatic reaction and baby's medical risk. Infant Behav Dev. 2007 Dec;30(4):679-84. doi: 10.1016/j.infbeh.2007.03.004. Epub 2007 Apr 20. PMID 17449102
- [Background] DeBoer RW, Karemaker JM, Strackee J. Comparing spectra of a series of point events particularly for heart rate variability data. IEEE Trans Biomed Eng. 1984 Apr;31(4):384-7. doi: 10.1109/TBME.1984.325351. No abstract available. PMID 6745974
- [Background] Hofer MA. Early social relationships: a psychobiologist's view. Child Dev. 1987 Jun;58(3):633-47. PMID 3608643
- [Background] Als H, Lawhon G, Duffy FH, McAnulty GB, Gibes-Grossman R, Blickman JG. Individualized developmental care for the very low-birth-weight preterm infant. Medical and neurofunctional effects. JAMA. 1994 Sep 21;272(11):853-8. PMID 8078162
- [Derived] Welch MG, Barone JL, Porges SW, Hane AA, Kwon KY, Ludwig RJ, Stark RI, Surman AL, Kolacz J, Myers MM. Family nurture intervention in the NICU increases autonomic regulation in mothers and children at 4-5 years of age: Follow-up results from a randomized controlled trial. PLoS One. 2020 Aug 4;15(8):e0236930. doi: 10.1371/journal.pone.0236930. eCollection 2020. PMID 32750063
- [Derived] Beebe B, Myers MM, Lee SH, Lange A, Ewing J, Rubinchik N, Andrews H, Austin J, Hane A, Margolis AE, Hofer M, Ludwig RJ, Welch MG. Family nurture intervention for preterm infants facilitates positive mother-infant face-to-face engagement at 4 months. Dev Psychol. 2018 Nov;54(11):2016-2031. doi: 10.1037/dev0000557. Epub 2018 Oct 4. PMID 30284883
- [Derived] Hane AA, Myers MM, Hofer MA, Ludwig RJ, Halperin MS, Austin J, Glickstein SB, Welch MG. Family nurture intervention improves the quality of maternal caregiving in the neonatal intensive care unit: evidence from a randomized controlled trial. J Dev Behav Pediatr. 2015 Apr;36(3):188-96. doi: 10.1097/DBP.0000000000000148. PMID 25757070
- [Derived] Welch MG, Hofer MA, Stark RI, Andrews HF, Austin J, Glickstein SB, Ludwig RJ, Myers MM; FNI Trial Group. Randomized controlled trial of Family Nurture Intervention in the NICU: assessments of length of stay, feasibility and safety. BMC Pediatr. 2013 Sep 24;13:148. doi: 10.1186/1471-2431-13-148. PMID 24063360
- [Derived] Welch MG, Hofer MA, Brunelli SA, Stark RI, Andrews HF, Austin J, Myers MM; Family Nurture Intervention (FNI) Trial Group. Family nurture intervention (FNI): methods and treatment protocol of a randomized controlled trial in the NICU. BMC Pediatr. 2012 Feb 7;12:14. doi: 10.1186/1471-2431-12-14. Erratum In: BMC Pediatr. 2012;12:107. PMID 22314029